CLINICAL TRIAL: NCT00003042
Title: Dose-Intense Chemotherapy and Stem Cell Rescue in the Treatment of Inflammatory Breast Carcinoma
Brief Title: Chemotherapy and Stem Cell Transplantation in Treating Patients With Stage IIIB Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 96139; P30CA033572 (NIH); CHNMC-96139; NCI-G97-1288; CDR0000065672 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: stage IIIB breast cancer; inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Filgrastim; Cisplatin; Cyclophosphamide; Doxorubicin; Melphalan; Mesna; Paclitaxel; Tamoxifen; Peripheral Blood Stem Cell Transplantation

ARMS (2):
- 1 cycle of neoadjuvant chemotherapy (Experimental): Patients receive chemotherapy, surgical removal of the cancer followed by additional chemotherapy, followed by two treatment cycles of very high-dose chemotherapy, return of bone marrow derived cells, followed by radiation therapy and if indicated five years of tamoxifen treatment.
  Interventions: Biological: filgrastim; Drug: cisplatin; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: melphalan; Drug: mesna; Drug: paclitaxel; Drug: tamoxifen citrate; Procedure: bone marrow ablation with stem cell support; Procedure: conventional surgery; Procedure: peripheral blood stem cell transplantation
- More than 1 cycle of neoadjuvant chemotherapy (Experimental): Patients receive chemotherapy, followed by two treatment cycles of very high-dose chemotherapy, return of bone marrow derived cells, followed by radiation therapy and if indicated five years of tamoxifen treatment.
  Interventions: Biological: filgrastim; Drug: cisplatin; Drug: doxorubicin hydrochloride; Drug: melphalan; Drug: mesna; Drug: paclitaxel; Drug: tamoxifen citrate; Procedure: bone marrow ablation with stem cell support; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: cisplatin
Drug: cyclophosphamide
  Arms: 1 cycle of neoadjuvant chemotherapy
Drug: doxorubicin hydrochloride
Drug: melphalan
Drug: mesna
Drug: paclitaxel
Drug: tamoxifen citrate
Procedure: bone marrow ablation with stem cell support
Procedure: conventional surgery
  Arms: 1 cycle of neoadjuvant chemotherapy
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: This phase II trial is studying how well chemotherapy and stem cell transplantation work in treating patients with stage IIIB breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effectiveness of neoadjuvant dose intensive sequential chemotherapy, followed by surgical resection, adjuvant therapy, and tandem high dose chemotherapy and stem cell rescue in patients with inflammatory stage IIIB breast cancer.
* Determine the clinical and pathological remission rate (complete, partial, and overall) following neoadjuvant dose dependent sequential chemotherapy in patients with inflammatory stage IIIB breast cancer.
* Determine the relapse and survival rate of these patients with the above therapy.
* Determine the potential correlations between inflammatory features and hereditary background.

OUTLINE: Patients are stratified according to those who have had no more than 1 cycle of neoadjuvant chemotherapy (stratum 1) and those who have had more than 1 cycle of neoadjuvant chemotherapy and/or modified radical mastectomy (stratum 2).

Patients in stratum 1 receive doxorubicin IV over 96 hours on days 1-4, 15-19, and 29-32. Paclitaxel is infused over 96 hours on days 43-47 and 57-60. Filgrastim (G-CSF) is administered on days 5-10, 20-25, 33-38, 48-55, and 61-68, and beyond if the granulocyte count is less than 1000/mm^3. A modified radical mastectomy is performed between days 70 and 80. All stratum 1 and stratum 2 patients then receive paclitaxel IV for 96 hours on days 100-104, and cyclophosphamide IV on day 121. Filgrastim is administered at one dose on days 105-110 and days 122-127 and at a higher dose on days 110-116 and days 128-135. Stem cells are harvested from the patient on days 113-116 and days 132-135.

High-dose chemotherapy is then administered to all patients in the study. Course 1 starts with doxorubicin IV on days -7 to -3. Paclitaxel IV is administered for 24 hours on day -2. Filgrastim is administered by IV on day -1 and continued until the granulocyte count is greater than 1000/mm^3 for 3 days. Peripheral stem cells are reinfused on day 0. Course 2 starts 4-6 weeks after the start of course 1 with melphalan and cisplatin being infused on day -11. Filgrastim is administered IV on days -10 to -6. Melphalan and cisplatin are administered again on day -4. Stem cells are infused on day -3 and on day 0. Filgrastim is then administered until the granulocyte count is at least 1000/mm^3 for 3 days.

Radiation therapy is started 4-7 weeks after the beginning of course 2. Tamoxifen is started within 2 weeks of discharge following course 2 in patients with hormone receptor positive tumors.

Patients are followed every 3 months for two years and then annually for the next three years.

PROJECTED ACCRUAL: Approximately 60 patients will be accrued, at a rate of about 15 per year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage IIIB breast cancer with dermal/epidermal invasion or clinical features of inflammation, erythema, pain or hypersensitivity, edema, or thickening of the skin
* Diagnosis within the past 6 months

PATIENT CHARACTERISTICS:

Age:

* 60 and under

Performance status:

* Karnofsky 80-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 mg/dL
* SGOT or SGPT no greater than 1.5 times the upper limit of normal

Renal:

* Creatinine less than 1.2 mg/dL
* Creatinine clearance at least 80 mL/min
* No history of hemorrhagic cystitis

Cardiovascular:

* Left ventricular fraction at least 55% on MUGA scan
* No previous valvular heart disease or arrhythmia

Pulmonary:

* FEV_1 at least 60% predicted
* Room air pO_2 greater than 85 mmHg
* Room air pCO_2 no greater than 43 mmHg
* DLCO at least 60% of the lower limit of predicted value

Other:

* No history of malignant disease in the past 5 years, except for squamous or basal cell skin cancer and stage I or in situ cervical cancer
* No organic CNS dysfunction
* Not pregnant
* No known and potentially disabling psychosocial history
* Not positive for hepatitis B or HIV

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Stratum 1:

  * No more than one cycle of chemotherapy
* Stratum 2:

  * No greater than 225 mg/m^2 doxorubicin and no greater than 250 mg/m^2 paclitaxel during previous chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiation to the left chest wall

Surgery:

* Modified radical mastectomy allowed

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 1997-05-30 (Actual); Primary Completion 2010-02-09 (Actual); Study Completion 2025-12-29 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: George Somlo, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Neoadjuvant Chemo Followed by Surgery & High-dose Chemo With PSC Rescue: Patients receive chemotherapy, surgical removal of the cancer followed by additional chemotherapy, followed by two treatment cycles of very high-dose chemotherapy, return of bone marrow derived cells, followed by radiation therapy and if indicated five years of tamoxifen treatment.
  filgrastim
  cisplatin
  cyclophosphamide
  doxorubicin hydrochloride
  melphalan
  mesna
  paclitaxel
  tamoxifen citrate
  bone marrow ablation with stem cell support
  conventional surgery
  peripheral blood stem cell transplantation
- High-dose Chemo With Rescue: Following surgery patients receive chemotherapy, followed by two treatment cycles of very high-dose chemotherapy, return of bone marrow derived cells, followed by radiation therapy and if indicated five years of tamoxifen treatment.
  filgrastim
  cisplatin
  doxorubicin hydrochloride
  melphalan
  mesna
  paclitaxel
  tamoxifen citrate
  bone marrow ablation with stem cell support
  peripheral blood stem cell transplantation
Period: Overall Study
Arm/Group | Neoadjuvant Chemo Followed by Surgery & High-dose Chemo With PSC Rescue | High-dose Chemo With Rescue
Started | 14 | 27
Completed | 14 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neoadjuvant Chemo Followed by Surgery & High-dose Chemo With PSC Rescue | High-dose Chemo With Rescue | Total
Number analyzed (Participants) | 14 | 27 | 41
Age, Continuous [Median (Full Range); unit: years] | 49 [30 to 61] | 50 [34 to 61] | 50 [30 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 27 | 41
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13 | 25 | 38
  Hispanic | 1 | 1 | 2
  Black | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 27 | 41

OUTCOME MEASURES:

1. Primary Outcome: Three-year Relapse-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Relapse defined as appearance of any new lesions during or after protocol treatment.
Time Frame: From date of mastectomy until date of relapse or death from any cause, 3 years post mastectomy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neoadjuvant Chemo Followed by Surgery & High-dose Chemo With PSC Rescue | High-dose Chemo With Rescue
Number analyzed (Participants) | 14 | 27
percentage of participants | 61.5 [30.8 to 81.8] | 77.8 [57.1 to 89.3]

2. Primary Outcome: Five-year Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Endpoint is defined as death due to any cause.
Time Frame: From date of mastectomy until date of death, 5 years post mastectomy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neoadjuvant Chemo Followed by Surgery & High-dose Chemo With PSC Rescue | High-dose Chemo With Rescue
Number analyzed (Participants) | 14 | 27
percentage of participants | 69.2 [37.3 to 87.2] | 70.4 [49.4 to 83.9]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed during all cycles of chemotherapy treatment (up to 6 months).
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Neoadjuvant Chemo Followed by Surgery & High-dose Chemo With PSC Rescue | High-dose Chemo With Rescue
All-Cause Mortality (participants affected / at risk) | 10/14 | 14/27
Serious Adverse Events (participants affected / at risk) | 0/14 | 2/27
Other Adverse Events (participants affected / at risk) | 13/14 | 23/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Chemo Followed by Surgery & High-dose Chemo With PSC Rescue (N=14) | High-dose Chemo With Rescue (N=27)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Chemo Followed by Surgery & High-dose Chemo With PSC Rescue (N=14) | High-dose Chemo With Rescue (N=27)
Cerebellar (Nervous system disorders) | 4 (7) | 10 (19)
Dysrhythmias (Cardiac disorders) | 4 (8) | 9 (15)
Fluid Retention (Renal and urinary disorders) | 5 (24) | 10 (26)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 6 (25) | 11 (27)
Ischemia (Cardiac disorders) | 4 (8) | 9 (15)
Pericardial (Cardiac disorders) | 4 (8) | 9 (15)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 5 (24) | 10 (26)
Stomatitis (General disorders) | 5 (24) | 10 (26)
Weight (Food Intake) (Metabolism and nutrition disorders) | 5 (16) | 9 (9)
Clinical Coagulation (Blood and lymphatic system disorders) | 2 (2) | 7 (12)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (6) | 11 (15)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 3 (5)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
EF/CHF (Cardiac disorders) | 4 (8) | 9 (15)
Left ventricular failure (Cardiac disorders) | 3 (4) | 4 (4)
Myocardial ischemia (Cardiac disorders) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 5 (7) | 10 (13)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hearing (Ear and labyrinth disorders) | 4 (7) | 10 (16)
Hearing loss (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vision (Eye disorders) | 4 (7) | 10 (19)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 8 (9)
Constipation (Gastrointestinal disorders) | 5 (16) | 18 (30)
Diarrhea (Gastrointestinal disorders) | 6 (18) | 13 (25)
Diarrhea (Somlo COH) (Gastrointestinal disorders) | 2 (2) | 7 (10)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia, esophagitis, odynophagia (Somlo COH) (Gastrointestinal disorders) | 1 (1) | 1 (2)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (6) | 3 (4)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incontinence NOS (Gastrointestinal disorders) | 2 (2) | 2 (3)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 3 (4)
Nausea (Gastrointestinal disorders) | 10 (26) | 18 (34)
Nausea (Somlo COH) (Gastrointestinal disorders) | 2 (2) | 7 (11)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Stomatitis/phayngitis (Somlo COH) (Gastrointestinal disorders) | 2 (2) | 7 (10)
Vomiting (Gastrointestinal disorders) | 10 (25) | 19 (35)
Vomiting (Somlo COH) (Gastrointestinal disorders) | 1 (1) | 7 (11)
Chest pain (General disorders) | 1 (1) | 5 (5)
Chills (General disorders) | 3 (4) | 9 (9)
Fatigue (General disorders) | 8 (14) | 8 (11)
Fever (General disorders) | 2 (4) | 5 (6)
Fever (no infection) (General disorders) | 4 (11) | 10 (21)
General symptom (General disorders) | 2 (2) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 4 (5)
Irritability (General disorders) | 1 (2) | 0 (0)
Oedema NOS (General disorders) | 5 (6) | 11 (14)
Pain (General disorders) | 4 (7) | 8 (12)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1) | 1 (1)
Allergy (Immune system disorders) | 5 (24) | 10 (26)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Catheter related infection (Infections and infestations) | 1 (1) | 3 (3)
Infection, Bacterial (COH) (Infections and infestations) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
AGC (Investigations) | 5 (20) | 10 (25)
Activated partial thromboplastin time prolonged (Investigations) | 5 (6) | 10 (15)
Alanine aminotransferase increased (Investigations) | 1 (2) | 5 (6)
Alk Phos (Somlo COH) (Investigations) | 1 (1) | 1 (1)
Alkaline Phosphatase (Investigations) | 4 (8) | 7 (7)
Alkaline phosphatase increased (Investigations) | 2 (4) | 5 (7)
Amylase (Investigations) | 3 (5) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Bilirubin (Investigations) | 4 (8) | 7 (7)
Bilirubin (Somlo COH) (Investigations) | 1 (1) | 0 (0)
Creatinine (Investigations) | 2 (2) | 3 (3)
Creatinine increased (Investigations) | 3 (3) | 4 (5)
HGB/HCT (Investigations) | 4 (13) | 8 (8)
Hyperbilirubinemia (Investigations) | 0 (0) | 1 (1)
Hypercholesterolemia (Investigations) | 0 (0) | 1 (1)
INR increased (Investigations) | 6 (8) | 13 (17)
Leukopenia (Investigations) | 1 (1) | 1 (1)
Lymphopenia (Investigations) | 0 (0) | 2 (4)
Neutrophil count decreased (Investigations) | 3 (6) | 3 (6)
Neutrophils (ANC) (Somlo COH) (Investigations) | 3 (5) | 8 (14)
(Investigations) | 7 (39) | 9 (53)
Partial Thromboplastin Time (Investigations) | 2 (2) | 7 (11)
Platelet count decreased (Investigations) | 2 (4) | 5 (8)
Platelets (Investigations) | 5 (20) | 10 (25)
Platelets (Somlo COH) (Investigations) | 3 (4) | 8 (14)
Prothrombin Time (Investigations) | 2 (2) | 7 (12)
SGOT (Somlo COH) (Investigations) | 1 (1) | 0 (0)
SGOT/SGT (Investigations) | 4 (8) | 7 (7)
SGPT (Somlo COH) (Investigations) | 0 (0) | 2 (2)
WBC (Investigations) | 4 (13) | 8 (8)
Weight gain (Investigations) | 3 (4) | 3 (3)
Weight loss (Investigations) | 1 (2) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 4 (5) | 9 (14)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (10) | 10 (22)
Hyperglycemia (Metabolism and nutrition disorders) | 12 (24) | 23 (43)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 12 (22) | 22 (42)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (10) | 10 (22)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 10 (17) | 21 (37)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (6)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Cortical/State of Consciousness (Nervous system disorders) | 4 (7) | 11 (20)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 5 (5)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 10 (15) | 17 (29)
Motor Activity (Nervous system disorders) | 4 (7) | 10 (19)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (2)
Neurological disorder NOS (Nervous system disorders) | 2 (3) | 1 (1)
Peripheral Nervous System Sensory (Nervous system disorders) | 4 (7) | 10 (19)
Peripheral motor neuropathy (Nervous system disorders) | 3 (4) | 7 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (9) | 12 (19)
Speech disorder (Nervous system disorders) | 1 (2) | 1 (1)
Taste alteration (Nervous system disorders) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 4 (7) | 7 (7)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 6 (7)
Hallucination NOS (Psychiatric disorders) | 0 (0) | 2 (2)
Ideation (Psychiatric disorders) | 4 (7) | 10 (19)
Insomnia (Psychiatric disorders) | 3 (4) | 5 (5)
Mood (Psychiatric disorders) | 4 (7) | 10 (19)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0)
Blood urine present (Renal and urinary disorders) | 3 (3) | 2 (2)
Hematuria (Renal and urinary disorders) | 2 (2) | 3 (3)
Proteinuria (Renal and urinary disorders) | 2 (2) | 3 (3)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 6 (7)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 5 (5)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (12) | 9 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Extensive Skin Rash (Skin and subcutaneous tissue disorders) | 2 (5) | 7 (9)
Local Skin Rash (Skin and subcutaneous tissue disorders) | 2 (5) | 7 (9)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (2) | 5 (7)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 5 (9) | 6 (7)
Sweating (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 3 (3) | 3 (3)
Hemorrhage (Vascular disorders) | 7 (26) | 13 (29)
Hypertension (Vascular disorders) | 5 (6) | 17 (23)
Hypotension (Vascular disorders) | 7 (8) | 17 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT00003042/Prot_SAP_000.pdf